CLINICAL TRIAL: NCT02520258
Title: Study of the Reversibility of Glucose Intolerance Caused by Chronic Aspartame Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Thomas Huber, Research Assistant Professor, Rockefeller University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: THU-0887
Record Dates: First submitted 2015-07-30; First posted 2015-08-11 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Glucose Metabolism Disorder
Keywords: artificial sweeteners; obesity; diabetes; metabolic syndrome; aspartame
MeSH Terms: conditions — Glucose Metabolism Disorders; Obesity; Diabetes Mellitus; Metabolic Syndrome | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspartame Consumers - Cohort 1 (Experimental): Experimental Group/Arm
  Phase I - Questionnaires and fasting oral glucose tolerance test (OGTT).
  Phase II - (If OGTT results are abnormal, participants will be invited to participate in Phase II) Five (5) week study phase with Prudent Metabolic Diet and Intervention of diet soda containing aspartame only; Week 1: Prudent Metabolic Diet and 36oz diet soda po daily, Week 2-4: Prudent Metabolic Diet and no diet soda, Week 5: Prudent Metabolic Diet and 36 oz diet soda po daily.
  Interventions: Other: Oral glucose tolerance test (OGTT); Other: Diet soda containing aspartame only
- Aspartame Naive Participants - Cohort 2 (Active Comparator): Control Group/Arm
  Phase I - Questionnaires and fasting oral glucose tolerance test (OGTT).
  Phase II - Not applicable for this cohort.
  Interventions: Other: Oral glucose tolerance test (OGTT)

INTERVENTIONS:
Other: Oral glucose tolerance test (OGTT) — OGTT will be conducted following a ten (10) hour fast on Screening Visit 2 (Screening Visit 2 may be conducted between Day -42 to Day 1).
Other: Diet soda containing aspartame only — 7 days of 36 oz diet soda po daily (Week 1), followed by 21 days washout (Weeks 2-4), and 7 days rechallenge (Week 5); Prudent metabolic diet; Oral glucose tolerance test (OGTT) on days (+/-2) 3, 7, 10, 14, 21, 28, 31, 35
  Arms: Aspartame Consumers - Cohort 1

SUMMARY:
Experiments have shown that some artificial sweeteners like those in diet soda can cause changes in how the body responds to and uses sugar. These changes increase the chance of obesity, type 2 diabetes, and other metabolic diseases. In this study, the investigators plan to see if the most common artificial sweetener, aspartame (brand name Equal, NutraSweet), causes these changes. The investigators believe that if metabolic changes are observed in a person who consumes aspartame, then removing all aspartame from the diet might lead to a reversal of the changes and a normalization of test results.This would impact sweetener additives in our foods and thus decrease the incidence of obesity, diabetes, and the metabolic syndrome.

DETAILED DESCRIPTION:
Experiments have shown that some artificial sweeteners like those in diet soda can cause changes in how the body responds to and uses sugar. These changes increase the chance of obesity, type 2 diabetes mellitus, and other metabolic diseases. In this study, the investigators plan to see if the most commonly used artificial sweetener, aspartame, affects the body's response to sugar. The investigators believe that if metabolic changes are observed in a person who consumes aspartame, then removing all aspartame from the diet might lead to a reversal of the changes and a normalization of test results.

The investigators plan to study two (2) cohorts of healthy volunteers: 1) Those who regularly drink at least three cans per day of diet soda that contains aspartame (Cohort 1, Aspartame Consumers) and 2) participants who consume less than or equal to two (2) cans of diet soda per week (Cohort 2, Aspartame Naïve Participants).

Phase I of the study, the investigators will ask participants questions about their usual diet, including how much diet soda they usually drink. Participants will be screened by a test called the oral glucose tolerance test, or OGTT. This test involves coming to the hospital to drink sugary syrup, then have blood sugar checked every thirty (30) minutes for five (5) hours. Before the test, participants must refrain from eating or drinking anything for ten (10) hours. If the OGTT shows a high value, then the participant in cohort 1 (Aspartame Consumers) who regularly drink 3 or more cans per day of diet soda will be approached about continuing into the second phase of the study. For the participants in cohort 2 (consume less than or equal to two (2) cans of diet soda per week; Aspartame Naïve Participants), this will be the end of their participation in the study.

Phase II of the study, blood tests, OGTT, stool samples, and weight and body fat measurements a few times a week will track any changes in the participants during the study. During the phase II five (5) week study, participants will receive all of their meals from the Rockefeller University Hospital and should not have any outside food or drinks. The diet used throughout this study phase (II) is the Prudent Metabolic Diet. Participants can leave the hospital and continue to work, but must come for all tests and to receive meals. During Week One, participants will eat only food provided by the hospital but will continue to drink three (3) cans of diet soda per day. In Weeks Two through Four, participants will continue to eat food given to them by the hospital and will not be allowed to consume any foods or drinks that contain aspartame. In Week Five, participants will continue on the hospital diet, but will again start drinking three (3) cans of diet soda per day.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 - 45
2. Weight stable for at least 3 months prior to screening (< 5% weight change)
3. BMI of 21 - 29
4. Cohort 1 - Aspartame Consumers: Primary dietary sweetener is aspartame; consumes at least 36 ounces of diet soda in which aspartame is a primary ingredient (Diet Coke or Diet Dr Pepper) a day for at least 6 months duration prior to study enrollment (Primary dietary sweetener is aspartame" should be defined as: "840g per week sucrose equivalent from aspartame and less than 280 grams per week sucrose equivalent from all other sweeteners (non-caloric and caloric sweeteners). For reference, one 12oz soda is 40g sucrose equivalent, and one teaspoon (one packet) of artificial sweetener is 4g sucrose equivalent.)"

   Cohort 2 - Aspartame Naïve Participants: Consumes less than or equal to 2 cans of diet soda per week
5. Screening Visit #2 OGTT Outcome:

   * 0-h plasma glucose < 110 mg/dl AND
   * 2-h plasma glucose < 140 mg/dl
6. Abnormal OGTT during the screening phase of the study (area under curve on the high end of distribution)
7. Must be able to comply with a metabolic Prudent diet
8. Willing to fast 10 hours before each OGTT and BodPod
9. Current level of exercise (aerobic and/or resistance training) must be able to be sustained while an in-patient

Exclusion Criteria:

1. Any evidence of US National Cholesterol Education Program Adult Treatment Panel III

   Clinical Identification of the Metabolic Syndrome (must have 3 or more of the following risk factors):

   Abdominal Obesity, given as a waist circumference:
   * Men >102 cm (>40 in)
   * Women > 88 cm (>35 in)

   Triglycerides >150 mg/dl

   HDL Cholesterol:
   * Men < 40 mg/dl
   * Women <50 mg/dl

   Blood Pressure >130/ >85 mm Hg

   Fasting Glucose > 110 mg/dl
2. Average systolic blood pressure (SBP) > 150 mmHg and / or diastolic blood pressure (DBP) > 90 mmHG (based on 3 BPs taken at screening visit #1),
3. LDL-C > 240mg/dl
4. Triglycerides > 400 mg/dl
5. Evidence of a liver disorder (ALT > three fold of the ULN)
6. Evidence of any renal disease
7. Currently on a weight-loss diet
8. Diabetes
9. Self-reported history of thyroid dysfunction
10. Sugar sweetened beverage consumption (> 84 ounces per week)
11. Hemoglobin <13.0 g/dl for males and 12.0 g/dl for females
12. Current, prior (within 2 months), or anticipated use of any of the following medications:

    antihyperlipidemic, hyperglycemic medications, Antineoplastics, Antiretrovirals, Selective Serotonin Reuptake Inhibitors, Diuretics, Antihypertensives, Anticonvulsants, Hormone therapy, Birth control
13. Self-reported antibiotic use within the previous 3 months
14. Currently pregnant or lactating
15. History of cardiac disease
16. Active illegal drug user (self-reported)
17. History of GI surgery (gastric bypass, bariatric, Roux-en-Y, colon resection, etc.)
18. Habitual ingestion of > 2 alcoholic beverages/day
19. Ever diagnosed with an eating disorder (self-reported)
20. Use of steroids or beta agonists (orally, intranasal or inhaled) within a week of any OGTT
21. Positive Hepatitis Serology (Hep. B surface Antibody; Hep. B surface antigen; Hep. C surface antibody)
22. HIV Positive
23. Tobacco use within the past 3 months
24. Any medical or social condition that, in the opinion of the Investigator, might pose additional risk to the participant or confound the results of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Interval changes in blood glucose | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in blood glucose will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Blood glucose | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): Blood glucose will be quantified from incremental area under the curve calculated from averaged oral glucose tolerance tests (OGTT)

SECONDARY OUTCOMES:
Interval changes in Glucagon | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in glucagon will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Glucagon | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): glucagon will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)
Interval changes in Peptide Tyrosine Tyrosine (PYY) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in PYY will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Peptide Tyrosine Tyrosine (PYY) | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): PYY will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)
Interval changes in Leptin | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in Leptin will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Leptin | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): Leptin will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)
Interval changes in Insulin | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in Insulin will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Insulin | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): Insulin will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)
Interval changes in Ghrelin | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in Ghrelin will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Ghrelin | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): Ghrelin will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)
Interval changes in Glucagon-like peptide-1 (GLP-1) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in GLP-1 will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Glucagon-like peptide-1 (GLP-1) | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): GLP-1 will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)
Interval changes in Glucose-dependent insulin-releasing peptide (GIP) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in GIP will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
Glucose-dependent insulin-releasing peptide (GIP) | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): GIP will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)
Interval Changes in C-peptide | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  Phase II (cohort 1): Interval changes in C-peptide will be quantified from area under the curve calculated from oral glucose tolerance tests (OGTT)
C-peptide | Screening Visit 2: conducted between day -42 up to Day 1.
  Phase I (both cohorts): C-peptide will be quantified from area under the curve calculated from averaged oral glucose tolerance tests (OGTT)

OTHER OUTCOMES:
Interval changes in glycated hemoglobin (HbA1C) - Phase II (Cohort 1) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
Glycated hemoglobin (HbA1C) - Phase I (both cohorts) | Screening Visit 2: conducted between day -42 up to Day 1.
Interval changes in body mass index (BMI) - Phase II (Cohort 1) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
  BMI is calculated from measured height and weight
Body mass index (BMI) - Phase I (both cohorts) | Screening Visit 2: conducted between day -42 up to Day 1.
  BMI is calculated from measured height and weight
Interval changes in body fat distribution - Phase II (Cohort 1) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
Body fat distribution - Phase I (both cohorts) | Screening Visit 2: conducted between day -42 up to Day 1.
Interval changes in whole body densitometry (BodPod) - Phase II (Cohort 1) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
Whole body densitometry (BodPod) - Phase I (both cohorts) | Screening Visit 2: conducted between day -42 up to Day 1.
Interval changes in blood pressure - Phase II (Cohort 1) | Interval 1: days 1 to 7; interval 2: days 8 to 28; interval 3: days 29 to 35
Blood pressure - Phase I (both cohorts) | Screening Visit 2: conducted between day -42 up to Day 1.
Interval changes in frequency distribution of microbes found in stool samples (Phase II - cohort 1) | Interval 1: days 6 to 7; interval 2: days 27 to 28; interval 3: days 34 or 35.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Huber, MD PhD, Principal Investigator — Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No